CLINICAL TRIAL: NCT03645655
Title: PIVKA-II Combined With Alpha-Fetoprotein for Diagnostic and Prognostic Value of Hepatic Tumors in Infants: Protocol for a Multicenter, Observational Study
Brief Title: PIVKA-II Combined With Alpha-Fetoprotein for Diagnostic and Prognostic Value of Hepatic Tumors in Infants
Acronym: PIVKA-II
Status: Completed | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Chidren's Hospital of Fudan University (Unknown); Chongqing Children's Hospital, Chongqing Medical University (Unknown); Children's Hospital of Nanjing Medical University (Other); Qilu Children's Hospital of Shandong University (Other); Anhui Children's Hospital (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Zhengzhou Children's Hospital (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: General surgery of SCMC
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Hepatoblastoma; Hepatic Hemangioendothelioma
Keywords: hepatoblastoma; Hepatic Hemangioendothelioma; Protein induced by vitamin K absence or antagonist-II; Alpha-fetoprotein; infant; Differential diagnosis
MeSH Terms: conditions — Hepatoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood was collected from each patient prior to any treatment (surgery and/or chemotherapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hepatoblastoma: The diagnosis of hepatoblastoma is based on enhanced CT scanning and/or histopathology.
  Interventions: Diagnostic Test: PIVKA-II
- hepatic hemangioendothelioma: The diagnosis of hepatic hemangioendothelioma is based on enhanced CT scanning and/or histopathology.
  Interventions: Diagnostic Test: PIVKA-II
- Healthy control: The healthy control group consist of people undergoing routine medical examination.

INTERVENTIONS:
Diagnostic Test: PIVKA-II — Serum samples are tested for tumor markers including PIVKA-II, AFP, and biochemical tests.
  Other Names: DCP
  Groups: hepatic hemangioendothelioma; hepatoblastoma

SUMMARY:
Although hepatic tumors are uncommon in the perinatal period they are associated with significant morbidity and mortality in affected patients. The study is intended to evaluate the diagnostic efficiency of Protein Induced by Vitamin K Absence or antagonist-II(PIVKA-II) combining with alpha-fetoprotein in hepatic tumor of infant. This study is a multicenter study joined by several hospitals in China. Participants including hepatoblastoma, hepatic hemangioendothelioma and healthy control are consecutively recruited into the cohort. All the serum samples are collected before and after each treatment and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II, alpha-fetoprotein and biochemical indexes including alanine aminotransferase(ALT), aspartate aminotransferase(AST), gamma-glutamyl transferase(GGT), alpha-l-fucosidase(AFU), etc.

DETAILED DESCRIPTION:
Hepatic tumors seldom occur in the perinatal period. They comprise approximately 5% of the total neoplasms of various types occurring in the fetus and neonate. Infantile hemangioendothelioma is the leading primary hepatic tumor followed by hepatoblastoma. Although alpha-fetoprotein has been well recognized as biomarker of hepatic tumors, it should be mentioned that this protein in normal infants is highly elevated during the first 2 months of life.

Protein induced by vitamin K antagonist-II (PIVKA-II), also known as des-γ-carboxyprothrombin (DCP) or acarboxy prothrombin, is an abnormal form of prothrombin induced by vitamin K absence or antagonist-II. An elevated serum level of PIVKA-II is reported to be associated with hepatocellular (HCC). Many studies have shown that PIVKA-II is applicable for HCC surveillance and has been written into the guideline of JSH, which achieves remarkably good results.

The study is intended to evaluate diagnostic and differential diagnostic accuracy of PIVKA-II combining with alpha-fetoprotein in hepatic tumor of infant.

This study is a multicenter study joined by several hospitals in China. Participants including hepatoblastoma, hepatic hemangioendothelioma and healthy control. All the serum samples are collected before and after each treatment and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II, Alpha-fetoprotein(AFP)， and biochemical indexes including ALT, AST, GGT, AFU, etc. The diagnosis of hepatoblastoma and hepatic hemangioendothelioma was based on enhanced CT scanning and/or histopathology. The Student's t-test (or Mann-Whitney test) was used to compare continuous variables, and the chi-square test (or Fisher's exact test) was used for categorical variables. A receiver operator characteristic (ROC) curve was used to assess the diagnostic and differential diagnostic efficiency of PIVKA-II and the combined tumor markers with AFP.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 12 month
* Receiving no treatment before diagnosis
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Serum samples doesn't qualified
* Vitamin K absence

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will be recruited through inpatient department.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change of PIVKA-II | Baseline Time, Postoperative Day 1
  Using PIVKA-II assay kit (ARCHITECT I2000SR REFURB, Abbott, America).

SECONDARY OUTCOMES:
Change of AFP | Baseline Time, Postoperative Day 1
  Using the AFP assay (ARCHITECT AFP, Abbott, America).

CONTACTS AND LOCATIONS:
Overall Officials: Min Xu, Doctor, Study Chair — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao H, Xie C, Wang J, Ma J, Liu S, Xie L, Zheng Y, Dong R, Wang S, Fang Y, Wu Y, Zhang X, Lu X, Li Y, Li W, Pan Q, Xu M, Gu S. PIVKA-II combined with alpha-fetoprotein for the diagnostic value of hepatic tumors in children: a multicenter, prospective observational study. Hepatol Int. 2024 Aug;18(4):1326-1335. doi: 10.1007/s12072-024-10668-4. Epub 2024 Apr 16. PMID 38622445